CLINICAL TRIAL: NCT04622306
Title: A Randomized, Masked, 3-way Cross-over, Multi-center, Clinical Investigation to Evaluate Two Polyurethane Condoms in Healthy Monogamous Couples Compared With a Standard Latex Condom
Brief Title: Evaluation of Polyurethane Male Condoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sagami Rubber Industries Co., Ltd. (Industry)
Collaborators: Essential Access Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: SAGCS 2; NCT05763264 (obsolete NCT alias)
Record Dates: First submitted 2020-11-02; First posted 2020-11-09 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Contraception; Prevention of Sexually Transmitted Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Control Latex Condom C (Active Comparator): Commercial Natural Rubber Latex Male Condom
  Interventions: Device: Control Latex Condom C, Polyurethane Condom A, Polyurethane Condom B
- Polyurethane Condom A (Experimental): Polyurethane Condom A (002)
  Interventions: Device: Control Latex Condom C, Polyurethane Condom A, Polyurethane Condom B
- Polyurethane Condom B (Experimental): Polyurethane Condom B (001)
  Interventions: Device: Control Latex Condom C, Polyurethane Condom A, Polyurethane Condom B

INTERVENTIONS:
Device: Control Latex Condom C, Polyurethane Condom A, Polyurethane Condom B — Condom functionality study to determine failure rates

SUMMARY:
The clinical study will compare two lubricated polyurethane male condoms of different thickness with a marketed lubricated control male condom made of natural rubber latex. This crossover study will randomize 300 heterosexual couples to the sequence in which they use five condoms of each of the three study condom types. The clinical failure (breakage and slippage) rates of the two polyurethane condoms will be compared to the clinical failure (breakage and slippage) rate of commercial natural rubber latex control condom using a statistical test of non-inferiority. The study will also compare the acceptability of the two polyurethane condom different thickness with that of the natural rubber latex control condom obtained from interviews and questionnaires with subject couples.

DETAILED DESCRIPTION:
The clinical study will compare two lubricated polyurethane male condoms of different thickness and different sizes with a marketed lubricated control male condom made of natural rubber latex.

Couples entering the study will be expected to use 5 of each type of the 3 condoms in a randomised order. The identity of the condoms will be masked to both the couples and the investigators. The aim will be to recruit 300 heterosexual with the intent of achieving a minimum 1,000 uses of each condom type. Couples will report condom use events using a condom report form. The primary information collected will relate to condom breakage and slippage of the penis during use.

The total clinical failure rates (breakage and slippage) of the two polyurethane condoms will be compared to the clinical failure (breakage and slippage) rate of commercial natural rubber latex control condom using a statistical test of non-inferiority. The study will also compare the acceptability of the two polyurethane condom different thickness with that of the natural rubber latex control condom obtained from interviews and questionnaires with subject couples.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 45 (inclusive)
2. Protected against pregnancy by oral contraceptives, an IUD, an implant, contraceptive injections, contraceptive patch, or sterilization (tubal ligation or vasectomy)
3. Have home internet access, a valid personal email for each partner, ability to videoconference and use electronic signature technology
4. Willing and able to give electronic informed consent
5. Willing to respond to questions concerning their reproductive and contraceptive history and use of condoms via interview or self-administered questionnaires
6. Have vaginal intercourse at least once weekly
7. Willing to use the study products for fifteen acts of vaginal intercourse within nine weeks of study entry
8. In a mutually exclusive monogamous relationship with their study partner for at least 6 months and be willing to remain mutually monogamous throughout study participation
9. Both study partners have previous experience using male condoms
10. Agree not to use any additional vaginal or sexual lubricant except the AstroglideTM product provided, if desired, supplied by the study
11. Agree not to expose the study condoms to jewelry (hand, facial, or genital) or piercings (facial or genital) that could damage the study condoms.
12. Agree not to use sex toys or drugs intended to enhance or diminish sexual response when using study condoms
13. Male partner agrees to ejaculate during vaginal intercourse
14. Agree to (or partner) hold the condom at the base of the erect penis during withdrawal
15. Agree to return any condoms that break during use
16. Agree to return any unopened condoms
17. Reachable by telephone

Exclusion Criteria:

1. Currently participating in another similar clinical study
2. Female partner self-reported as pregnant
3. Allergic to natural rubber latex or polyurethane, or has a history of recurrent adverse events following use of latex or polyurethane products
4. Unable to follow study requirements, use instructions or attend study visits or exchanges
5. Have a significant (high) risk of STIs, including HIV infection, or having a medical history of recurrent, uncontrolled STIs (e.g. gonorrhoea, syphilis, Chlamydia, etc.)
6. Currently using condoms for protection against a known STI
7. Taking any internally applied medication to treat a genital condition that could interact with the study condom
8. Male partner has used medication that has caused erectile dysfunction, or had difficulty achieving/maintaining an erection, or achieving ejaculation in the last month under typical circumstances/conditions
9. Male has had a prostatectomy
10. Any self-reported genitourinary condition (e.g. itching, burning, irritation, etc.) which, in the opinion of the investigator, could affect use of the study condoms or the ability to interpret study data
11. Employee or affiliate of Essential Access Health or Sagami Rubber Industries Co., Ltd.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant R Burt, Study Chair — Sagami Rubber Industries Co., Ltd.; William D Potter, PhD, Study Director — Stapleford Scientific Services Limited
Locations (1):
- Essential Access Health, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Potter W, Burt G, Walsh T. Clinical breakage, slippage and acceptability of two commercial ultra-thin polyurethane male condoms compared to a commercial thin latex condom: a randomised, masked, 3 way crossover, multi centre controlled study (SAGCS 2). Reprod Health. 2024 Sep 4;21(1):128. doi: 10.1186/s12978-024-01873-3. PMID 39232840

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The total recruitment target was 300 couples consented couples (600 participants). Each couple to participate in each of the 6 arms using 5 condoms of each type in a randomized block sequence. The six randomized sequences were ABC, ACB, BAC, BCA, CAB, CBA.
  Each couple received 5 of the first assigned condom at the start of the study along with a set of 5 blank condom reports. Couples also received a penis measuring kit.
  The couples were expected to use all 15 condoms within 9 weeks.
Groups:
- Couples Assigned to Sequence ABC: Couples assigned at random to use the condoms in order Condom A first followed by Condom B then Condom C.
- Couples Assigned to Sequence ACB: Couples assigned at random to use the condoms in order Condom A first followed by Condom C then Condom B.
- Couples Assigned to Sequence BAC: Couples assigned at random to use the condoms in order Condom B first followed by Condom A then Condom C.
- Couples Assigned to Sequence BCA: Couples assigned at random to use the condoms in order Condom B first followed by Condom C then Condom A.
- Couples Assigned to Sequence CAB: Couples assigned at random to use the condoms in order Condom C first followed by Condom A then Condom B.
- Couples Assigned to Sequence CBA: Couples assigned at random to use the condoms in order Condom C first followed by Condom B then Condom A.
Period: Couples Used First Assigned Condom Set
Arm/Group | Couples Assigned to Sequence ABC | Couples Assigned to Sequence ACB | Couples Assigned to Sequence BAC | Couples Assigned to Sequence BCA | Couples Assigned to Sequence CAB | Couples Assigned to Sequence CBA
Started | 48 | 50 | 48 | 51 | 53 | 50
Completed | 46 (Condoms remaining at the end of the period were not used or were used in violation of the protocol.) | 48 | 48 | 51 | 51 | 45
Not Completed | 2 | 2 | 0 | 0 | 2 | 5
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0 | 2 | 5
Period: Couples Used Second Assigned Condom Set
Arm/Group | Couples Assigned to Sequence ABC | Couples Assigned to Sequence ACB | Couples Assigned to Sequence BAC | Couples Assigned to Sequence BCA | Couples Assigned to Sequence CAB | Couples Assigned to Sequence CBA
Started (Couples received their second randomly assigned set of 5 condoms along with 5 blank report forms.) | 46 | 48 | 48 | 51 | 51 | 45
Completed | 46 (Condoms remaining at the end of the period were not used or were used in violation of the protocol.) | 48 | 48 | 51 | 51 | 45
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Couples Used Third Assigned Condom Set
Arm/Group | Couples Assigned to Sequence ABC | Couples Assigned to Sequence ACB | Couples Assigned to Sequence BAC | Couples Assigned to Sequence BCA | Couples Assigned to Sequence CAB | Couples Assigned to Sequence CBA
Started (Couples received their third set of randomly assigned set of 5 condoms and blank report forms.) | 46 | 48 | 48 | 51 | 51 | 45
Completed | 46 (Condoms remaining at the end of the period were not used or were used in violation of the protocol.) | 48 | 46 | 48 | 51 | 45
Not Completed | 0 | 0 | 2 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is the number of couples who were consented to join the study
Groups:
- Overall Study Population: The total number of couples consented was 300 (600 participants). These were randomly assigned to the 6 arms of the study.
Arm/Group | Overall Study Population
Number analyzed (Participants) | 600
Age, Categorical [Count of Participants; unit: Participants] — Population: The participants were recruited as monogamous sexually active couples. The total recruited populated consisted therefore of 300 men and 300 women.
  Participants
    Male: number analyzed (Participants) | 300
    Male: <=18 years | 0
    Male: Between 18 and 65 years | 300
    Male: >=65 years | 0
    Female: number analyzed (Participants) | 300
    Female: <=18 years | 0
    Female: Between 18 and 65 years | 300
    Female: >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 300
  Male | 300
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Number recruited: Hispanic or Latino | 144
  Number recruited: Not Hispanic or Latino | 456
  Number recruited: Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 600
Number of participants completing study as per protocol [Count of Participants; unit: Participants] | 568

OUTCOME MEASURES:

1. Primary Outcome: Non Inferiority Analysis of Each of the Experimental Condoms Verses the Control Condom With Respect to Clinical Failure Rates (Combined Breakage and Slippage) as Per ISO 29943-1:2017.
Description: To confirm each experimental condom is non-inferior to the control condom with respect to total clinical failure rate. The definition of total clinical failure rate as specified in ISO 29943-1:2017 will be used. The Total Clinical Failure Rate is Defined as the Number of Condoms with at least One Acute Failure Event (e.g. Clinical Breakage or Clinical Slippage) Divided by the Number of Condoms Used During Intercourse; Typically Reported as a Percentage; Any Condom which Experiences Multiple Clinical Failure Events Only Count as a Single Clinical Failure.
  To be eligible for inclusion in the non-inferiority analysis the each couple had to have used at least one of the appropriate experimental condoms and at least one control condom. This means that the numbers of participants and condoms reported in each of the two non-inferiority comparisons will differ.
Time Frame: Self Completion of Questionnaires Within 12 Hours of condom use. Questionnaires returned to investigators when receiving next set of 5 condoms. All sets of questionnaires returned within 9 weeks of couple starting.
Population: The number of participants and condoms used for the non-inferiority assessment of Condom A versus Condom C and the equivalent numbers in the non-inferiority assessment of Condom B versus Condom C differ because some men found Condom B to be too small to use.
Measure: Count of Units; unit: Condom uses
Units Other Than Participants: Condom uses
Groups:
- Polyurethane Condoms A Used in Non-inferiority Analysis Condom A of Versus Condom C: The number of participants using Condom A included in the non-inferiority analysis of Polyurethane Condom A versus Control Latex Condom C.
- Latex Condoms C Used in Non-inferiority Analysis of Condom A Versus Condom C: The number of participants using Control Latex Condom C included in the non-inferiority analysis of Polyurethane Condom A versus Control Latex Condom C.
- Polyurethane Condoms B Used in Non-inferiority Analysis of Condom B Versus Condom C: The number of participants using Condom B included in the non-inferiority analysis of Polyurethane Condom A versus Control Latex Condom C.
- Latex Condom C Used in Non-inferiority Analysis of Condom B Versus Condom C: The number of participants using Control Condom C included in the non-inferiority analysis of Polyurethane Condom B versus Control Latex Condom C.
Arm/Group | Polyurethane Condoms A Used in Non-inferiority Analysis Condom A of Versus Condom C | Latex Condoms C Used in Non-inferiority Analysis of Condom A Versus Condom C | Polyurethane Condoms B Used in Non-inferiority Analysis of Condom B Versus Condom C | Latex Condom C Used in Non-inferiority Analysis of Condom B Versus Condom C
Number analyzed (Participants) | 504 | 504 | 494 | 494
Number analyzed (Condom uses) | 1193 | 1212 | 1142 | 1193
Condom uses
  Primary Analysis of Study Data: Clinical Breaks | 15 | 10 | 22 | 9
  Primary Analysis of Study Data: Clinical slippages | 13 | 6 | 13 | 6
  Primary Analysis of Study Data: Successful Uses | 1165 | 1196 | 1107 | 1178
  Post hoc Analysis of Condom B versus Condom C where male penis length limited to ≤ 170 mm.: number analyzed (Participants) | 0 | 0 | 380 | 380
  Post hoc Analysis of Condom B versus Condom C where male penis length limited to ≤ 170 mm.: number analyzed (Condom uses) | 0 | 0 | 886 | 915
  Post hoc Analysis of Condom B versus Condom C where male penis length limited to ≤ 170 mm.: Clinical Breaks | 0 | 0 | 12 | 5
  Post hoc Analysis of Condom B versus Condom C where male penis length limited to ≤ 170 mm.: Clinical slippages | 0 | 0 | 8 | 6
  Post hoc Analysis of Condom B versus Condom C where male penis length limited to ≤ 170 mm.: Successful Uses | 0 | 0 | 866 | 904
Statistical Analysis 1: Comparison: Polyurethane Condoms A Used in Non-inferiority Analysis Condom A of Versus Condom C vs Latex Condoms C Used in Non-inferiority Analysis of Condom A Versus Condom C; Null Hypothesis: Expected test condom total clinical failure rate - expected control natural rubber latex male condom total clinical failure rate ≥ δ, where δ = 2.5%; Power calculations were conducted according to ISO 29943-1:2017. Target sample sizes were chosen to provide a power of at least 90%; Test type: Non-Inferiority — The non-inferiority margin for the difference in total clinical failure rates (clinical breakage plus clinical slippage) between the test and control condom is specified in ISO 23409:2011 as 2.5%; p = 0.025, GEE — The p-value was adjusted to 0.025 since two comparisons are being made on the data set; Upper 97.5% CL for difference = 2.5, 97.5% CI 1-sided [upper limit 2.5]
Statistical Analysis 2: Comparison: Polyurethane Condoms B Used in Non-inferiority Analysis of Condom B Versus Condom C vs Latex Condom C Used in Non-inferiority Analysis of Condom B Versus Condom C; Null Hypothesis: Test condom total clinical failure rate - control natural rubber latex male condom total clinical failure rate ≥ δ, where δ = 2.5%; Power calculations were conducted according to ISO 29943-1:2017. Target sample sizes were chosen to provide a power of at least 90%; Test type: Non-Inferiority — The non-inferiority margin for the difference in total failure rates (clinical breakage plus clinical slippage) between the test and control condom is specified on ISO 23409:2011 as 2.5%; p = 0.025, GEE — The p-value was adjusted to 0.025 since two comparisons are being made on the data set; Upper 97.5% CLof difference = 2.5, 97.5% CI 1-sided [upper limit 2.5]
Statistical Analysis 3: Comparison: Polyurethane Condoms B Used in Non-inferiority Analysis of Condom B Versus Condom C vs Latex Condom C Used in Non-inferiority Analysis of Condom B Versus Condom C; The non-inferiority analysis was repeated after removing couples where the male partner had a penis length greater than 170 mm. The polyurethane condom B has a specified nominal length of 170 mm and is not recommended for men with penises longer than the length of the condom; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p = 0.025, GEE — The p-value was adjusted to 0.025 since two comparisons are being made on the data set; Upper 97.5% CL for difference = 2.37, 97.5% CI 1-sided [upper limit 2.5]

ADVERSE EVENTS:
Time Frame: Participants completed report forms after each condom use. Each condom report elicited information about specific adverse event usually experienced when using condoms including discomfort caused by burning, irritation and itching sensations, rashes, constriction, decreased sensitivity and dryness. Participants were expected to use all 15 condoms within 9 weeks, which can therefore be regarded as the monitoring period for adverse event.
Description: All adverse events were rated by severity (mild, moderate, severe), duration (only while wearing condom, 1 to 10 minutes after condom removed, 11 to 59 minutes after condom removed and more than 59 minutes after condom removed.
Arm/Group | Polyurethane Condom A | Polyurethane Condom B | Control Latex Condom C
All-Cause Mortality (participants affected / at risk) | 0/337 | 0/392 | 0/332
Serious Adverse Events (participants affected / at risk) | 4/337 | 10/392 | 20/332
Other Adverse Events (participants affected / at risk) | 41/337 | 85/392 | 87/332
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polyurethane Condom A (N=337) | Polyurethane Condom B (N=392) | Control Latex Condom C (N=332)
Discomfort caused by irritation, burning sensation, itching or rash (Skin and subcutaneous tissue disorders) | 4 (4) | 10 (10) | 20 (20)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polyurethane Condom A (N=337) | Polyurethane Condom B (N=392) | Control Latex Condom C (N=332)
Mild to moderate discomfort (Skin and subcutaneous tissue disorders) | 41 (41) | 85 (85) | 87 (87) — Causes of mild to moderate discomfort include burning, irritation, itching, rash, constriction, decreased sensitivity and dryness.

LIMITATIONS AND CAVEATS:
All condom use events were self reported. There is a potential for misreporting the number of events.

Since the trial was masked it was not feasible to preselect men with smaller penises to use the smaller Condom B. Instead, a post hoc analysis of the association between penis size and clinical failure rates was conducted followed by a further non-inferiority analysis after excluding men with penis lengths exceeding the specified nominal length of Condom B (170 mm).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT04622306/Prot_SAP_000.pdf